CLINICAL TRIAL: NCT02045654
Title: Retrospective Study for Predictive Marker for Decitabine Treament in MDS Patients
Brief Title: Platelet Response During the Second Cycle of Decitabine Can Predict Response and Survival for Myelodysplastic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jun Ho Jang, Professor, Samsung Medical Center
Other Study IDs: 2014-01-086
Record Dates: First submitted 2014-01-15; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDS patients: MDS patients who were treated with decitabine

SUMMARY:
To assess the efficacy of decitabine and identify predictors for response to decitabine therapy.

DETAILED DESCRIPTION:
* Histologically confirmed Myelodysplastic syndrome Diagnosed with MDS (de novo or secondary) based on the World Health Organization (WHO) classifications
* Survival and response Analysis
* Response rate
* Overall survival
* Leukemia free survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Myelodysplastic syndrome Diagnosed with MDS (de novo or secondary) based on the World Health Organization (WHO) classifications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed Myelodysplastic syndrome Diagnosed with MDS (de novo or secondary) based on the World Health Organization (WHO) classifications
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-02 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Response rate | 1 year
  International Working Group (IWG) response criteria

SECONDARY OUTCOMES:
Overall survival | 1 year
  measured from the date of decitabine therapy to the date of death or the last follow-up visit
Leukemia free survival | 1 year
  the date of decitabine therapy to the date of death or leukemic transformation

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Jang, Pf, Principal Investigator — Samsung Medical Center
Locations (1):
- Division of Hematology Oncology, Samsung Medical Center, Seoul, South Korea